CLINICAL TRIAL: NCT07083999
Title: Prospective Observational Study to Evaluate Fertility in Women Between 32 and 38 Years Old Treated With the Ovosicare® Fertility Food Supplement Containing a Combination of MYO/DCI in a 3.6:1 Ratio, Antioxidants, Vitamins and Minerals
Brief Title: Observational Study to Evaluate Fertility in Women Between 32 and 38 Years Old Treated With the Ovosicare® Fertility
Acronym: FERTILOBS
Status: Recruiting | Type: Observational
Sponsor: Procare Health Iberia S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: FERTILOBS
Record Dates: First submitted 2025-02-07; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Fertility
Keywords: FERTILOBS; Pregnancy; Food supplement; Ovosicare Fertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Suplementation: Women on Ovosicare Fertility supplementation prescribed according to standard clinical practice

SUMMARY:
The goal of this observational study is to evaluate whether supplementation with the Ovosicare® Fertility food supplement increases the possibility of becoming pregnant in women aged between 32 and 38 years who have been trying to become pregnant for at least 6 months before starting supplementation.

DETAILED DESCRIPTION:
The duration of participation in the study for each patient will be a maximum of 18 months. This follow-up period may be shorter if a pregnancy occurs.

The number of visits throughout the study will be a total of three. Please note that you will not have to undergo additional tests or attend any extraordinary visits due to participating in this study, since the procedures you will undergo are the same as those routinely carried out in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. - Women who agree to participate in the study by signing the informed consent.
2. - Between 32 and 38 years old.
3. - Who come to doctor´s office stating that they have been trying to get pregnant for at least 6 months.

Exclusion Criteria:

1. - BMI > 30 kg/m2.
2. - Existence of severe male factor subfertility according to the criteria of the World Health Organization (WHO), with at least one analysis obtained in the last 6 months with one or more variables with values of:

   * Azoospermia
   * Progressive motility <25%
   * Normal morphology ≤2%
3. - Pregnant or breastfeeding women.
4. - Patients with type 1 diabetes or thyroid disease.
5. - Patients with any assisted reproduction technique scheduled during the duration of the study.
6. - Patients who have used or taken systemic steroids, anticonvulsants, antiretroviral treatment for HIV or hepatitis B in the last month.
7. - Patients with a known allergy to any of the components of Ovosicare® Fertility.
8. - Any other situation that, in the medical opinion, advises against treatment with Ovosicare® Fertility or that may make patient follow-up difficult.
9. - Patients with suspected endometriosis.
10. - Existence of fibroids affecting the endometrial cavity.
11. - Patients with 2 or more previous abortions.
12. - Patients with a current diagnosis of a high-risk human papillomavirus (HPV) cervical lesion.

Ages: 32 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study population will be approximately 300 women between 32 and 38 years of age who go to the doctor indicating that they are having difficulty getting pregnant (at least 6 months without getting pregnant), to whom a dietary supplement based on Myo-inositol and D-Chiro-inositol in combination (Ovosicare® Fertility) will be prescribed as per standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of spontaneous pregnancy in women between 32 and 38 years old after a maximum of 6 months of supplementation with Ovosicare Fertility | From enrollment to visit 2 (9 months)
  Women suspected of being pregnant will undergo a blood test to detect the hormone beta-hCG and a transvaginal ultrasound to confirm the pregnancy.

SECONDARY OUTCOMES:
Evaluate the time until spontaneous clinical pregnancy | From enrollment to visit 2 (9 months)
  The variable "time" (months) until pregnancy will be calculated using the following formula:
  Time (months)= (Date of pregnancy - Date of treatment intake) / 30.44
Evaluate changes in analytical parameters in blood: Biochemistry panel | From enrollment to visit 2 (9 months)
  Description: To evaluate physiological changes by measuring biochemistry levels in blood from patients who do not achieve spontaneous clinical pregnancy after 9 months from the start of supplementation.
Evaluate changes in analytical parameters in blood: Hormonal panel | From enrollment to visit 2 (9 months)
  To evaluate physiological changes by measuring hormonal levels in blood from patients who do not achieve spontaneous clinical pregnancy after 9 months from the start of supplementation.
Evaluate changes in karyotype | From enrollment to visit 2 (9 months)
  To evaluate changes in karyotype by measuring in blood from patients who do not achieve spontaneous clinical pregnancy after 9 months from the start of supplementation.
Evaluate the presence of anatomy changes by ultrasound test | From enrollment to visit 2 (9 months)
  To evaluate anatomic changes by ultrasound test in patients who do not achieve spontaneous clinical pregnancy after 9 months from the start of supplementation.
To evaluate changes in the number of antral follicle by ultrasound test | From enrollment to visit 2 (9 months)
  To evaluate changes in the number of antral follicle by ultrasound test in patients who do not achieve spontaneous clinical pregnancy after 9 months from the start of supplementation.
Evaluate the safety profile of Ovosicare Fertility | From enrollment to 6months (during sumplementation)
  The percentage of patients with adverse events (AE) and serious adverse events (SAE) wil be described, as well as the total number of AEs and SAEs recorded up to visit 2. AEs will be coded using the MedDRA dictionary and their characteristics will be described as qualitative variables in terms of severity, intensity, causal relationship, and assessment of the response.
Ovosicare Fertility tolerability degree | From enrollment to 6 months (during sumplementation)
  To evaluate the degree of tolerability of treatment with Ovosicare® Fertility by the investigator a qualitative variable will be collected considered as poor, bad, good, excellent.
Ovosicare Fertility use satisfaction degree | From enrollment to 6 months (during sumplementation)
  To evaluate the degree of investigator satisfaction with the use of Ovosicare® Fertility a qualitative variable will be collected considered as very insatisfied, insatisfied, satisfied, very satisfied
Ovosicare Fertility Adherence | From enrollment to 6 months (during sumplementation)
  Treatment adherence will be evaluated as a qualitative variable referring to the correct intake of treatment following the frequency prescribed by the investigator. The frequency is defined as: always, quite often, sometimes, never
Live birth rate | After 9 moths after pregnancy confirmation
  To evaluate the live birth rate

CONTACTS AND LOCATIONS:
Locations (27):
- Spain (27):
  - CM Sitges, Sitges, Barcelona
  - HU de Getafe, Getafe, Madrid
  - Clínica Rv Benalmádena, Benalmádena, Malaga
  - H García Orcoyen, Estella-Lizarra, Navarre
  - CP Dr. Andrade Andrade, A Coruña
  - CP Dra. Domenech Casanova, Alicante
  - H Vega Baja de Orihuela, Alicante
  - Clinica Alboran, Almería
  - CP Dr. Aragón Albillos, Almería
  - CM Teknon, Barcelona
  - CP Dra. Mallafre, Barcelona
  - HU Vall d'Hebron, Barcelona
  - OBS Ginecólogos Burgos, Burgos
  - Clínica Attella, Castelló
  - HU de Donostia, Donostia / San Sebastian
  - CP Dra. Skouri-Bnihech Tioua, Granada
  - CHU Insular - H Materno-Infantil, Las Palmas
  - Clínica Palacios, Madrid
  - Gymeiaka Dra. Oltra Badui, Madrid
  - Gymeiaka Dra. Pavón Sanz, Madrid
  - HU La Paz, Madrid
  - Clínica Imar, Murcia
  - Ancla Clínica Ginecológica, Pontevedra
  - HG de la Santísima Trinidad, Salamanca
  - CP Dra. Sánchez Quintana, Seville
  - HU i Politècnic la Fe, Valencia
  - Centro Ginecológico Bolonia, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided